CLINICAL TRIAL: NCT04211701
Title: Comparison of the Effects of Connective Tissue Massage and Classical Massage Methods on Pain, Flexibility, Disability and Autonomic Responses in Chronic Mechanical Back Pain, Randomized Study
Brief Title: Effects of Connective Tissue Massage and Classical Massage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2019-0177
Record Dates: First submitted 2019-11-25; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Body Temperature
Keywords: Connective Tissue; Massage; Peripheral Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective Tissue Massage (Experimental): Connective tissue massage will be applied to the lumbo-sacral region, lower thoracic, scapular and interscapular regions, respectively. The treatment will be administered for four weeks, five days a week.
  Interventions: Procedure: Connective Tissue Massage
- Classical Massage (Experimental): Classic massage will be applied to the lower back and upper back, respectively, while the patient is lying in the prone position. The treatment will be administered for four weeks, five days a week.
  Interventions: Procedure: Classical Massage

INTERVENTIONS:
Procedure: Connective Tissue Massage — Connective tissue massage (CTM) will be applied to the lumbo-sacral region, lower thoracic, scapular and interscapular regions. Three to five pulling will be applied during massage. The treatment will be administered for four weeks, five days a week.
  Arms: Connective Tissue Massage
Procedure: Classical Massage — Classic massage (CM) will be applied to the lower back and upper back while the patient is lying in the prone position. Three stroking will be applied during massage.The treatment will be administered for four weeks, five days a week.
  Arms: Classical Massage

SUMMARY:
As a randomized study, this study aimed to investigate the effects of classical massage and connective tissue massage on pain, flexibility, disability, quality of life and autonomic responses in patients with chronic mechanical low back pain. The primary evaluation parameter of the study is autonomic function and the secondary evaluation parameter is pain. The participants will be treated accompanied with same physiotherapist along four weeks and five days in a week. A six-week follow-up will be performed to see how long the effect of the treatment continues.

DETAILED DESCRIPTION:
Mechanical low back pain is defined as a condition that causes tension, pain, or stiffness in the lumbar region where it is not possible to define a specific cause (eg infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome or cauda equina syndrome). Low back pain has become one of the biggest problems for public health systems in the Western world in the second half of the 20th century and continues to be a major health problem worldwide today. In a review based on studies on low back pain in 54 countries, the prevalence of low back pain was found to be 18.3%. As a result of researches made in Turkey in the 18-24 age range prevalence of women was 28.9%, in men was 18.1%, with advanced age over the age of 55 rate increasing further, it raise 48.1% in women and 31.5% in men. As shown in the researches, low back pain is seen more frequently in the age of late 20s and in women.

Disc degeneration, nociceptive factors, tumor necrosis factor α and smoking have been reported to be reason in mechanical low back pain. Although there are widely used clinical tests for pathologies arising from lumbar structures (discogenic low back pain, facet joint pain, sacroiliac joint pain), these tests cannot be used to diagnose non-specific mechanical low back pain.

The affect of chronic pain on individuals is quite different. Pain creates problems in the life of the individual starting from minimal to high level of disability and consequently severely restricts their participation in work and social life and their roles in the family. Medicines used to reduce pain are addictive after a while. Therefore, researchers emphasized the need for more emphasis on non-pharmacological treatment approaches in the management of persistent low back pain. Among these approaches, manual treatment, exercise, massage, and acupuncture methods are included in the treatment guidelines for mechanical low back pain.

No method of treatment of low back pain can produce a permanent improvement. However, there are several approaches that reduce pain and disability. Among these, massage is considered as a safe treatment method due to its low side effects and risk. Massage has been shown to be effective in some types of headaches, post-exercise muscle pain, and mechanical neck pain, but is also reported to cause relaxation and psychological relaxation. Classical massage (CM) is thought to improve the physiological and clinical outcomes by providing symptomatic reduction in pain through physical and mental relief and by increasing pain threshold by endorphin release. It is also suggested that CM has some effects on the nervous system. Massage applications cause repetitive sensory stimulations to occur and changes in neuronal circuits, such as blood pressure, cause altered activity in the autonomic nervous system.

Connective tissue remodeling has been reported in patients with chronic low back pain due to emotional, behavioral and motor dysfunction. Increased stress due to excessive use, repetitive motion and / or hypermobility, and reduced stress due to immobilization or hypomobility, cause changes in the connective tissue. Chronic, local increase in stress can lead to micro-injury and inflammation, while the absence of stress in the tissue leads to connective tissue atrophy, architectural disorder, fibroses, adhesions and contractures.

Connective tissue massage (CTM), which is also included in the basic training of physiotherapy, is a technique developed in 1929. The effects of the technique are improvement in autonomic nervous system functions, increase in blood circulation, muscle relaxation, decrease in pain and increase in mobility. Autonomic nervous system is stimulated by cutaneo-visceral reflexes in the massage area. While increased sympathetic nervous system activity decreases with massage, the autonomic nervous system responses can be balanced by the increase in parasympathetic activity. Parasympathetic effect of vasodilatation and increase in blood flow in the vessels will accelerate the healing process and decrease in spasm and pain.

In the literature, CTM has been shown to be effective in fibromyalgia and neck pain. However, no study has been found regarding the results of CTM application in patients with chronic mechanical low back pain. Also the effects of both classical and connective tissue massage on local and peripheral circulation have not been studied sufficiently. The aim of this study is to determine the most effective manual treatment method by comparing the effects of classical massage and connective tissue massage on autonomic nervous system responses, pain, flexibility and disability, which will be applied in addition to the hot pillow and exercise treatments commonly used in the clinic of chronic mechanical low back pain.

Hypotheses:

H0: The effect of CTM and CM on pain is similar in individuals with chronic mechanical low back pain.

H1: The effect of CTM and CM on disability is similar in individuals with chronic mechanical low back pain.

H2: The effect of CTM and CM applications on flexibility is similar in individuals with chronic mechanical low back pain.

H3: The effect of CTM and CM on autonomic functions is similar in individuals with chronic mechanical low back pain.

Material and Method:

The study will be conducted on individuals diagnosed with chronic mechanical low back pain by specialist physician. Individuals who meet the inclusion and exclusion criteria and sign the informed consent form will be randomly divided into two different groups by minimization method. One group will be treated with CTM (CTM Group) and the other with classical massage (CM Group).

In order to determine the number of individuals to be included in the study, power analysis was performed with GPower 3.0 program. As a result of the calculation using Cohen d: 0.8 α: 0.05, β: 0.2 (for 80% power) with the double-legged Mann-Whitney U test, it was found that 27 individuals would be needed each group and total of 54 individuals should be taken for trial. Considering that 30% of the individuals cannot comply with the treatment protocols to be applied (for reasons of time etc.), our sample size was increased by 30% and 35 individuals for each group were decided to have a final sample size of 70 people.

Individuals will be assess pain, disability, flexibility and autonomic functions before the treatment begins, after all treatments are complete and six weeks after treatment. In addition, the severity of pain will be measured every week during the treatment process, and pain and autonomic functions will be assess at the 20th treatment to see the acute effect of the treatment method.

Assessments:

Socio-Demographic Information Form: Information about the age, gender, height, body weight, occupation and background of the individuals will be recorded.

Pain Severity Measurement: Pain level of the individuals will be measured using the Visual Analogue Scale (VAS). The pain measurement will be performed before the start of treatment, at the end of the last treatment each week, 15 minutes after the session in the 20th treatment to see the acute effect of the treatment, after all treatments are finished and six weeks after the treatments are finished.

Assessment of Disability: In the assessment of disability due to low back pain, the Oswestry Low Back Pain Questionnaire will be used. The measurements will take place before the start of treatment and at the end of all treatment sessions and six weeks after the end of treatment.

Health Related Quality of Life Measurement: The Turkish version of the Short Form-36 (SF-36) questionnaire will be used to assess the quality of life related to health. The measurements will take place before the start of treatment, at the end of all treatment sessions and six weeks after the end of treatment.

Flexibility Measurements: Sit and reach test and lumbar lateral flexion measurements will be used to evaluate the lumbar flexibility of individuals. Measurements will take place before the start of treatment and at the end of all treatment sessions and six weeks after treatment is finished.

Sit and Reach Test: Individuals taking part in the test will sit on the floor with their bare feet, knees in extension, with the soles of the feet fully in contact with the test table. The part where the feet coincide on the test table shall be accepted as zero point and the tape measure shall be placed beyond and beyond this point. Values ahead from the zero point will be recorded as positive and the behind of the zero will be recorded as negative. The person will be asked to reach slowly on the test table with his hands flat and parallel to the floor and the upper extremities straight, the measured value from the end point of the fingers will be recorded in cm. The test will be performed twice and the average value will be recorded.

Lumbar Lateral Flexion Measurement: The individual will stand upright without shoes, with heels and back touching the wall and arms free. Before starting the test, the distance from the distal of the third finger to the floor will be measured with the help of tape measure and then the individual will be asked to flex his / her body to the lateral flexion without bending forwards or backwards and rotating and the distance between the distal of the third finger to floor will be measured again. The difference between the first measurement and the last measurement will be recorded. The measurement shall be made separately for the right and left sides. Within both sides, the test will be performed twice and the average value will be recorded.

Measurement of Autonomic Functions: Blood pressure, heart rate, peripheral temperature and local temperature changes will be measured to assess the effect of CTM and CM on possible autonomic responses in individuals. Measurements will be performed 30 minutes after these conditions if the individual is smoking or exercising. Heart rate will be measured with a pulse oximeter attached to the fingertip while the individual is sitting on the chair. To date, there has been no developed norm for peripheral temperature measurement. In the foot measurements using the thermogram, it was found that the hottest region on the plantar surface of the foot was the medial arch and the finger with the highest temperature was the first finger between the fingers. In line with the information obtained from these studies, measurements will be taken from the medial longitudinal arch. The environment in which the measurement is to be carried out is set at 25 °C and no direct sunlight and the individual will be asked to take off his shoes and socks and return to the supine position. It will be waited for 15 minutes for the moisture and temperature caused by the shoes and socks to disappear and return to normal temperature of the foot and then the measurement will be made with 'Testo' brand '830-T1 laser-marked heat meter.

In order to evaluate the effect of the applications on local heat, local temperature measurements will be made from the inferior corners of the ribs, from the top of the iliac crest and from the posterior superior iliac spine under the same laboratory environment and same conditions.

Peripheral and local temperature measurements will be performed before the start of treatment, 15 minutes after the end of the 20th treatment to measure the acute effect of the treatment method, after all treatments are finished and six weeks after the treatments are finished.

Interventions:

All participants will be treated with moist heat on the lumbar region for 20 minutes in all treatment sessions, followed by CTM in one group, CM in the other group and then exercise under the supervision of physiotherapist. Exercises will be combined with respiration with 10 repetitions. The exercise program will be:

Lumbar extensor muscle stretching in supine position (for 20 sec) Posterior pelvic tilt Bridging exercise Cat - camel exercise Hip twist - level 1 Clam - level 1

Connective Tissue Massage:

During CTM, individuals will be seated in a chair with the hip, knee and ankle at an angle of 90 degrees with all back and sacral regions open. It will be paid attention to the individual is slightly bent from the waist and the back is vertical. Hands will be supported on the thighs. Thus, a slight relaxation of the connective tissue will be achieved.

CTM will be applied to the lumbo-sacral area (basic section), lower thoracic region, scapular region and interscapular region respectively. In CTM, patients may experience normally expected sensations such as cutting and scratching, or a pathologically blunt feeling of pressure. Depth and number of repetitions will be increase or decrease according to individual's sense. In the CTM application, the distal phalanx of the third finger of the hand will be flexed to 45-60 degrees and short and long pulls will be made like hooking. Individuals will experience a feeling of shearing, scratching and blunt pressure due to therapist's pulling during the application. The speed of pulling will be increased or decreased according to the feeling of the individual. In the first 1-3 sessions of the application, the lumbo-sacral area will be taken and the pulling will be made to each field with 3-4 repetitions. Decreased tension and the appearance of hyperemia lines, the appropriate vascular response, will in turn be the criterion for progression to other regions. Approximately 3-4 sessions will be applied in other regions and an upper region will be added to the treatment when vascular reaction is obtained. Treatment sessions will start from five minutes to 20 - 25 minutes. CTM treatment will be continued for four weeks and a total of 20 sessions will be administered five times a week.

Classic Massage:

In classical massage application, lower back and upper back will be applied. The individual lies prone on treatment table in the inverted T position. Before starting the massage, massage oil will be applied to the application area and application will be started with the lower back area. Three general stroking respectively, followed by M. Erector spinae, M. Latissimus dorsi (first to the therapist's side, then opposite muscle), and M. gluteus maximus muscles three stroking, three kneading and three stroking respectively lower back application will be completed with general stroking.

After lower back massage, upper back massage will be started and no change will be made in the position of the individual. Following general stroking three times respectively during application, M. erector spinae and M. trapezius (first on the side of the therapist and then the opposite side) will be stroking three times, kneading three times and stroking three times, and general stroking will be completed three times and upper back application will be completed.

Classical massage will last for 15-20 minutes and will include five sessions per week and a total of 20 sessions with four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-60 years of age
* Low back pain for more than 12 weeks
* Lack of neurological problems caused by lumbar region
* Not to be included in physiotherapy and rehabilitation program in the last 6 months

Exclusion Criteria:

* Having ankylosing spondylitis
* Pain and / or numbness in the hip and lower extremities
* Previous trauma or surgery in lumbar region
* Presence of congenital malalignment in the vertebral column
* Malignancy
* Lower limb inequality over one cm
* Pregnancy
* Blood pressure difference of more than 10 mmHg between two arms

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2019-12-24 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Changes in autonomic function (pulse) compared with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about one minute.
  Pulse will be measured with pulse oximeter (pulse/min).
Changes in autonomic function (blood pressure) compared with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about two minutes
  Blood pressure will be measured with manual sphygmomanometer (mmHg).
Changes in autonomic function (temperature) compared with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about five minutes
  Local temperature and peripheral temperature measurements will be made with laser-marked heat meter (°C).
Changes in low back pain compared with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about one minute.
  Low back pain will be measured with using Visual Analog Scale (cm).

SECONDARY OUTCOMES:
Changes in disability compared to baseline with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about three minutes.
  Disability will be measured with Oswestry Disability Index (0 - 100)
Changes in quality of life compared to baseline with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about three minutes.
  Quality of life will be measured with Short Form 36 (0 - 100)
Changes in flexibility (lumbar lateral flexion test) compared to baseline with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about five minutes.
  Lumbar lateral flexion test will be measured with tape measure (cm).
Changes in flexibility (sit and reach) compared to baseline with baseline and last measurement | Measurements will be made at baseline and 4th week (last assessment). It takes about two minutes.
  Sit and reach test will be measured with special table (cm).
Changes in autonomic function (pulse) at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about one minute.
  Pulse will be measured with pulse oximeter (pulse/min).
Changes in autonomic function (blood pressure) at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about two minutes
  Blood pressure will be measured with manual sphygmomanometer (mmHg).
Changes in autonomic function (temperature) at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about five minutes
  Local temperature and peripheral temperature measurements will be made with laser-marked heat meter (°C).
Changes in low back pain at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about one minute.
  Low back pain will be measured with using Visual Analog Scale (cm)
Changes in disability at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about three minutes.
  Disability will be measured with Oswestry Disability Index (0 - 100)
Changes in quality of life at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about three minutes.
  Quality of life will be measured with Short Form 36 (0 - 100).
Changes in flexibility (lumbar lateral flexion) at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about two minutes.
  Lumbar lateral flexion test will be measured with tape measure (cm).
Changes in flexibility (sit and reach) at six weeks after the end of the treatment | Measurements will be made at six weeks after the end of the treatment. It takes about two minutes.
  Sit and reach test will be measured with special table (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Göktuğ Er, Principal Investigator — MPT; İnci Yüksel, Study Director — DPT
Locations (1):
- Eastern Mediterranean University, Mersin, Famagusta, Turkey (Türkiye)

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Oksuz E. Prevalence, risk factors, and preference-based health states of low back pain in a Turkish population. Spine (Phila Pa 1976). 2006 Dec 1;31(25):E968-72. doi: 10.1097/01.brs.0000247787.25382.3c. PMID 17139213
- [Background] Furlan AD, Imamura M, Dryden T, Irvin E. Massage for low back pain: an updated systematic review within the framework of the Cochrane Back Review Group. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1669-84. doi: 10.1097/BRS.0b013e3181ad7bd6. PMID 19561560
- [Background] Aourell M, Skoog M, Carleson J. Effects of Swedish massage on blood pressure. Complement Ther Clin Pract. 2005 Nov;11(4):242-6. doi: 10.1016/j.ctcp.2005.02.008. PMID 16290894
- [Background] Langevin HM, Sherman KJ. Pathophysiological model for chronic low back pain integrating connective tissue and nervous system mechanisms. Med Hypotheses. 2007;68(1):74-80. doi: 10.1016/j.mehy.2006.06.033. Epub 2006 Aug 21. PMID 16919887
- [Background] Kavlak E, Buker N, Altug F, Kitis A. Investigation of the effects of connective tissue mobilisation on quality of life and emotional status in healthy subjects. Afr J Tradit Complement Altern Med. 2014 Apr 3;11(3):160-5. doi: 10.4314/ajtcam.v11i3.23. eCollection 2014. PMID 25371578
- [Background] Yüksel İ, Baltacıoğlu S, Akbayrak T. Konnektif Doku Masajı. In: Yüksel İ, editor. Masaj Teknikleri. 4th ed. Ankara: Hipokrat Kitabevi & Pelikan Kitabevi; 2016. p. 283-354
- [Background] Bakar Y, Sertel M, Ozturk A, Yumin ET, Tatarli N, Ankarali H. Short term effects of classic massage compared to connective tissue massage on pressure pain threshold and muscle relaxation response in women with chronic neck pain: a preliminary study. J Manipulative Physiol Ther. 2014 Jul-Aug;37(6):415-21. doi: 10.1016/j.jmpt.2014.05.004. Epub 2014 Aug 6. PMID 25108749
- [Background] Holey LA, Dixon J, Selfe J. An exploratory thermographic investigation of the effects of connective tissue massage on autonomic function. J Manipulative Physiol Ther. 2011 Sep;34(7):457-62. doi: 10.1016/j.jmpt.2011.05.012. Epub 2011 Jul 23. PMID 21875520
- [Background] Toprak Celenay S, Anaforoglu Kulunkoglu B, Yasa ME, Sahbaz Pirincci C, Un Yildirim N, Kucuksahin O, Ugurlu FG, Akkus S. A comparison of the effects of exercises plus connective tissue massage to exercises alone in women with fibromyalgia syndrome: a randomized controlled trial. Rheumatol Int. 2017 Nov;37(11):1799-1806. doi: 10.1007/s00296-017-3805-3. Epub 2017 Aug 24. PMID 28840379
- [Background] Brattberg G. Connective tissue massage in the treatment of fibromyalgia. Eur J Pain. 1999 Jun;3(3):235-244. doi: 10.1053/eujp.1999.0123. PMID 10700351
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Koçyiğit H, Aydemir Ö, Ölmez N, Memiş A. Validity and reliability of Turkish version of Short form 36: A study of a patients with romatoid disorder. Drug and Therapy.1999; 12, 102-106
- [Background] Natour J, Cazotti Lde A, Ribeiro LH, Baptista AS, Jones A. Pilates improves pain, function and quality of life in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2015 Jan;29(1):59-68. doi: 10.1177/0269215514538981. Epub 2014 Jun 25. PMID 24965957
- [Background] Vischer AS, Burkard T. Principles of Blood Pressure Measurement - Current Techniques, Office vs Ambulatory Blood Pressure Measurement. Adv Exp Med Biol. 2017;956:85-96. doi: 10.1007/5584_2016_49. PMID 27417699
- [Background] Lahiri BB, Bagavathiappan S, Jayakumar T, Philip J. Medical applications of infrared thermography: A review. Infrared Phys Technol. 2012 Jul;55(4):221-235. doi: 10.1016/j.infrared.2012.03.007. Epub 2012 Apr 13. PMID 32288544
- [Background] Gatt A, Formosa C, Cassar K, Camilleri KP, De Raffaele C, Mizzi A, Azzopardi C, Mizzi S, Falzon O, Cristina S, Chockalingam N. Thermographic patterns of the upper and lower limbs: baseline data. Int J Vasc Med. 2015;2015:831369. doi: 10.1155/2015/831369. Epub 2015 Jan 13. PMID 25648145